CLINICAL TRIAL: NCT04367233
Title: Quadratus Lumborum Block Versus Transversus Abdominis Block . Randomized Clinical Trial.
Brief Title: Quadratus Lumborum Block Versus Transversus Abdominis Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Associate professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAAE 28763119.0.0000.5448
Record Dates: First submitted 2020-04-21; First posted 2020-04-29 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General

STUDY DESIGN:
Intervention Model Description: Prospective, controlled, randomized and double blinded.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A professional who will not participate in other stages of the study will conduct the drawing and envelopes preparation.
  Masking: at the end of the surgery, the anesthesiologist will perform the blocking corresponding to the patient's group and will not participate in other stages of the study. A professional who does not know the group to which each patient belongs will perform the collection and analysis of the endpoint variables.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Active Comparator): General anesthesia with fentanyl, propofol and remifentanyl
  Interventions: Other: General anesthesia
- Transverse block group (Experimental): At the end of general anesthesia with fentanyl, propofol and remifentanil, the patient will receive transverse plan block, with ropivacaine 0,25% 0,2 ml/kg.
  Interventions: Other: Transverse abdominal block
- Quadratus lumborum group (Experimental): At the end of general anesthesia with fentanyl, propofol and remifentanil, the patient will receive quadratus lumborum block with ropivacaine 0,25% 0,2 ml/kg.
  Interventions: Other: Quadratus lumborum block

INTERVENTIONS:
Other: General anesthesia — General anesthesia with fentanyl, propofol and remifentanil.
  Arms: Placebo group
Other: Transverse abdominal block — Transverse abdominal block with ropivacaine 0,25% 0,2 ml/kg at the end of general anesthesia with fentanyl, propofol and remifentanil
  Arms: Transverse block group
Other: Quadratus lumborum block — At the end of general anesthesia with fentanyl, propofol and remifentanil, patients will receive quadratus lumborum block with ropivacaine 0,25% 0,2 ml/kg
  Arms: Quadratus lumborum group

SUMMARY:
The advent of laparotomy replacement by minimally invasive techniques brought the obvious benefit of postoperative pain reduction. The application of transversus abdominis block has already demonstrated to reduce postoperative pain in laparoscopic hysterectomy. The comparison between it and quadratus lumborum block in cesarean sections showed that the latter was superior in relation to postoperative analgesia. The aim of this trial is to compare postoperative analgesia in patients receiving one or the other of these regional anesthesia techniques to prevent postoperative pain in gynecological laparoscopic surgeries. The recruited sample will be randomly distributed in three groups to receive placebo, transverse abdominal plan block or quadratus lumborum block, in a covert way for the patients and team. The primary outcome evaluated will be the postoperative consumption of opioid and the secondary outcome will be the evaluation of postoperative pain scores.

DETAILED DESCRIPTION:
: the sample will be divided into three groups and all participants will receive general anesthesia. Patients in the placebo group (PG) will be referred to the post-anesthesia recovery room after extubation and adequate hemodynamic and respiratory recovery. Patients in the tap block group (TBG) will receive 0.2 ml of 0.25% ropivacaine between the transverse and oblique internal muscles guided by ultrasound (US), on one side and after the other (the same dose), after the end of surgery. Patients in the quadratus lumborum group (LQG) will receive 0.2 ml/kg of 0.25% ropivacaine inside the middle layer of the thoracolumbar fascia guided by US, on one side and after the other (the same dose), after the end of the surgery. In all participants, the monitoring will include cardioscope, oximetry, non-invasive blood pressure and monitor of hypnoses level. After peripheral venous puncture, antibiotic prophylaxis with 2g cefazolin, and pre-anesthetic medication with midazolam 0.05 mg/kg. After 5 min pre-oxygenation, the patients will receive venous anesthetic induction with 2% lidocaine 1mg/kg without vasoconstrictor; fentanyl 4 µ/kg; propofol 2 mg/kg, or even adequate hypnosis guided by proper monitor; cisatracurium 0.15mg/kg, with tracheal intubation and mechanical ventilation after anesthetic plan confirmed with proper monitor and adequate muscle relaxation. Anesthesia will be maintained with propofol in continuous infusion guided by hypnoses monitor and remifentanil in continuous infusion between 0.1 and 0.5 µg/kg/min, according to patient need. All study participants will receive ondansetron 8 mg, dipyrone 2 g, ketoprofen 100 mg, dexamethasone 10 mg and morphine 3 mg. At the end of the surgery, after partial recovery from neuromuscular blockade, patients will receive atropine 0.01 mg/kg and neostigmine: 0.02mg/kg before tracheal extubation.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to gynecological video laparoscopy.

Exclusion Criteria:

* Allergy to any component of the study protocol, coagulopathies.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | 12 hours
  Consumption of morphine in the postoperative period,during hospital stay
Codeine consumption | Two days
  Consumption of codeine during the 48 hours following the surgery

SECONDARY OUTCOMES:
Postoperative pain | Two days
  Pain scores on awaking, 6 hours after, and during the first 2 postoperative days, based on verbal pain score, ranging 0 (without pain) to 10 (worst imaginable pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kelley WE Jr. The evolution of laparoscopy and the revolution in surgery in the decade of the 1990s. JSLS. 2008 Oct-Dec;12(4):351-7. No abstract available. PMID 19275847
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Suner ZC, Kalayci D, Sen O, Kaya M, Unver S, Oguz G. Postoperative analgesia after total abdominal hysterectomy: Is the transversus abdominis plane block effective? Niger J Clin Pract. 2019 Apr;22(4):478-484. doi: 10.4103/njcp.njcp_61_15. PMID 30975950
- [Background] Bacal V, Rana U, McIsaac DI, Chen I. Transversus Abdominis Plane Block for Post Hysterectomy Pain: A Systematic Review and Meta-Analysis. J Minim Invasive Gynecol. 2019 Jan;26(1):40-52. doi: 10.1016/j.jmig.2018.04.020. Epub 2018 Apr 30. PMID 29723644
- [Background] Verma K, Malawat A, Jethava D, Jethava DD. Comparison of transversus abdominis plane block and quadratus lumborum block for post-caesarean section analgesia: A randomised clinical trial. Indian J Anaesth. 2019 Oct;63(10):820-826. doi: 10.4103/ija.IJA_61_19. Epub 2019 Oct 10. PMID 31649394
- [Background] Ferreira KA, Teixeira MJ, Mendonza TR, Cleeland CS. Validation of brief pain inventory to Brazilian patients with pain. Support Care Cancer. 2011 Apr;19(4):505-11. doi: 10.1007/s00520-010-0844-7. Epub 2010 Mar 10. PMID 20221641